CLINICAL TRIAL: NCT05143073
Title: Understanding Genetic Risk for Alcohol Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HM20023103
Record Dates: First submitted 2021-11-19; First posted 2021-12-03 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Alcohol Use Disorder
Keywords: Genetic Feedback; Personalized Risk Information; Alcohol Use Disorder; Educational Intervention; Polygenic Risk Scores; Health Beliefs
MeSH Terms: conditions — Alcoholism; Genetic Risk Score | interventions — Ethanol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No educational materials (No Intervention): No educational materials will be provided.
- Alcohol use disorder and strategies to reduce risk (Active Comparator): The information provided to participants will be related to alcohol use disorder, including a definition, prevalence, consequences, risk factors, and risk-reducing strategies. The content is based on information from National Institute of Alcohol Abuse and Alcoholism websites, Mayo Clinic websites, and the National Survey on Drug Use and Health.
  Interventions: Behavioral: Alcohol use disorder and strategies to reduce risk educational material
- Complex polygenic risk scores, alcohol use disorder, and strategies to reduce risk (Active Comparator): The information provided to participants will explain polygenic risk scores by discussing genetic variation, risk variants, how polygenic scores are created, and how they can be interpreted. The participants will also receive the same information related to alcohol use disorder, including a definition, prevalence, consequences, risk factors, and risk-reducing strategies.
  Interventions: Behavioral: Complex polygenic risk scores, alcohol use disorder, and strategies to reduce risk educational material

INTERVENTIONS:
Behavioral: Alcohol use disorder and strategies to reduce risk educational material — Participants will be directed to educational information (~5 minutes) regarding alcohol use disorder and strategies to reduce risk which they will read.
  Arms: Alcohol use disorder and strategies to reduce risk
Behavioral: Complex polygenic risk scores, alcohol use disorder, and strategies to reduce risk educational material — Participants will be directed to educational information (~10 minutes) regarding complex polygenic risk scores, alcohol use disorder and strategies to reduce risk which they will read.
  Arms: Complex polygenic risk scores, alcohol use disorder, and strategies to reduce risk

SUMMARY:
The purpose of this study is to evaluate an online educational tool that will help individuals better understand alcohol use disorder, risk factors, and genetic risk information and to better understand participant's beliefs regarding alcohol use disorder. This study does not involve genetic testing. Investigators will not be giving participants any personalized genetic feedback as part of the study; however, investigators will ask participants to imagine that they receive different hypothetical genetic risk scores and respond to survey items.

DETAILED DESCRIPTION:
The purpose of this study is to conduct a randomized controlled trial to (1) evaluate the impact of receiving educational information about polygenic risk scores on an individual's ability to understand polygenic risk scores for alcohol use disorder, (2) assess the impact of receiving educational information about alcohol use disorder on components of behavior change theories including perceived severity of having alcohol problems, perceived benefits of taking actions to reduce risk for developing alcohol problems, and perceived barriers to taking risk reducing actions, and (3) assess how (hypothetical) genetic risk scores impact an individual's perceived chance of developing alcohol use disorder, future intentions, and an individual's psychological state.

The study aims to recruit 300 emerging adults from an urban, public university that will either be assigned to the control condition or one of two intervention groups. Participants in the intervention groups will either receive information about alcohol use disorder and ways to reduce risk or information about polygenic risk scores, alcohol use disorder, and ways to reduce risk. Emerging adults are the focus of this research proposal because they are entering a high-risk age range for the onset of many psychiatric conditions. Additionally, youth and young adults are high consumers of new technologies, with a majority using various digital technologies to access health information. Therefore, emerging adults may be more likely to access their genetic risk information as well as more likely to benefit from receiving genotypic information for alcohol use disorder, uniquely positioning emerging adults as the target population for this study.

Additionally, hypothetical genetic risk scores are provided to participants via three scenarios. Participants are asked to imagine they received each genetic risk score (low, average, high) and respond to a series of questions. The hypothetical genetic risk scores are provided using a graph based on the display of polygenic risk scores in the educational information. Low risk will be indicated using a graph in which the genetic risk score is in the 30th percentile, average risk will be indicated using a graph in which the genetic risk score is in the 50th percentile, and high risk will be indicated using a graph in which the genetic risk score is in the 75th percentile.

Outcomes from this research study are expected to contribute to our knowledge about how to provide genetic risk information for alcohol use disorder in a way to promote behavior change. The knowledge gained from the research will be critical to provide effective communication of genetic feedback for alcohol use disorder in the future in order to ensure results are delivered in a way that is beneficial to the individual, as well as inform policies and best practices regarding the return of personalized genetic feedback for alcohol use disorder and related psychiatric outcomes. Future research can build upon this knowledge by investigating the acute and long-term impact of returning actual genetic risk information for alcohol use disorder, which will further advance our understanding of the issues surrounding the return of complex genetic feedback.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate Virginia Commonwealth University students 18 or older
* Voluntary consent must be provided

Exclusion Criteria:

• Under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Understanding of genetic risk scores for alcohol use disorder | 1 hour
  Understanding of genetic risk scores for alcohol use disorder will be assessed after each of the three hypothetical scenarios in which participants receive a low genetic risk score, average genetic risk score, and high genetic risk score. Participants will respond to a series of true/false/don't know statements to assess understanding and interpretation of each genetic risk score. Responses will be scored as correct or incorrect and summed to create an overall score.
Perceived susceptibility of developing alcohol use disorder | 1 hour
  Perceived susceptibility for developing alcohol use disorder assesses an individual's belief about their chance of developing alcohol use disorder in the future. This will be measured using the Health Beliefs about Mental Illness Instrument. The items will be assessed immediately after the educational intervention and after each hypothetical genetic risk score. Five items from the Health Beliefs about Mental Illness Instrument will be scored from 1 (strongly disagree) to 5 (strongly agree) and averaged together to create an overall score.

SECONDARY OUTCOMES:
Perceived barriers to risk reducing behavior | 1 hour
  Perceived barriers to risk reducing behavior assesses perceived barriers to taking risk reducing actions which may include time, acceptability, and cost. This will be measured using the Health Beliefs about Mental Illness Instrument. Five items from the Health Beliefs about Mental Illness Instrument will be scored from 1 (strongly disagree) to 5 (strongly agree) and averaged together to create an overall score.
Perceived severity of alcohol use disorder | 1 hour
  Perceived severity of alcohol use disorder will assess beliefs about the severity of having alcohol problems on an individual's life. Perceived severity will be measured using the Health Beliefs about Mental Illness Instrument. Seven items from the Health Beliefs about Mental Illness Instrument will be scored from 1 (strongly disagree) to 5 (strongly agree) and averaged together to create an overall score.
Genetic knowledge | 1 hour
  Genetic knowledge related to psychiatric and substance use disorders will be assessed with an adapted version of the Public Understanding and Attitudes towards Genetics and Genomics Questionnaire (PUGGS). The PUGGS is an 11 item questionnaire which asks about the role of genetic and environmental risk factors in the development of substance use and psychiatric conditions. The number of correct answers is summed to yield a score ranging from 0 (very little understanding of genetic concepts related to psychiatric conditions) to 11 (high understanding of genetic concepts related to psychiatric conditions).
Future intentions | 1 hour
  Future intentions will assess whether the individual would seek additional information about alcohol use disorder, discuss risk with healthcare providers, believe it would be important to change drinking behavior, and intend to change drinking behaviors after receiving each hypothetical genetic risk score for alcohol use disorder. The response options for these items include yes, no, and unsure.
Hypothetical psychological impact of receiving a genetic risk score | 1 hour
  The hypothetical psychological impact of receiving a genetic risk score will be measured using an adapted version of the Impact of Event Scale. The adapted measure includes 10 items with responses scored from 1 (not at all) to 5 (extremely) which will be averaged to create an overall score. These items will be assessed in each hypothetical genetic risk scenario.
Self-perceived risk of developing alcohol use disorder | 1 hour
  Self-perceived risk of developing alcohol use disorder will be measured using an adapted item from Lipkus et al. 2015, a measure originally developed to assess perceived risk of nicotine addiction as a consequence of cigarette smoking. The item will be included immediately after the educational intervention and after each hypothetical genetic risk score. The self-perception of risk item adapted from Lipkus et al. 2015 will be coded as a semi-continuous variable from 1 (no chance) to 7 (certain to happen).
Worry about developing alcohol use disorder | 1 hour
  Worry about developing alcohol use disorder will be measured using an adapted version of the Cancer Worry Scale. Eight items from the adapted version of the Cancer Worry Scale will be scored from 1 to 4 and averaged together to create an overall score.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Dick, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Driver MN, Kuo SI, Dron JS, Austin J, Dick DM. The impact of receiving polygenic risk scores for alcohol use disorder on psychological distress, risk perception, and intentions to reduce drinking. Am J Med Genet B Neuropsychiatr Genet. 2023 Jul-Sep;192(5-6):93-101. doi: 10.1002/ajmg.b.32933. Epub 2023 Mar 1. PMID 36856135
- [Derived] Driver MN, Kuo SI, Petronio L, Brockman D, Dron JS, Austin J, Dick DM. Evaluating the impact of a new educational tool on understanding of polygenic risk scores for alcohol use disorder. Front Psychiatry. 2022 Nov 23;13:1025483. doi: 10.3389/fpsyt.2022.1025483. eCollection 2022. PMID 36506445